CLINICAL TRIAL: NCT04684810
Title: Lay Therapist Effectiveness With Displaced Persons Kurdish Iraq: Promising Exploratory Results for Global Mental Health Access
Brief Title: Lay Therapist Effectiveness With Displaced Persons Kurdish Iraq
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Meredith Blackwell, Principal Investigator, University of New Mexico
Other Study IDs: Jiyan01
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Mental Health; Therapeutics
Keywords: evidence-based treatments; refugee; lay therapists; global mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Group: Participants seeking treatment completed longitudinal data
  Interventions: Behavioral: Community Lay Therapist-Administered EBT

INTERVENTIONS:
Behavioral: Community Lay Therapist-Administered EBT — Community Therapists Used CBT and EMDR Interventions

SUMMARY:
Negative mental health effects of war exposure and displacement are pervasive, but many displaced persons and refugees in low-and-middle income countries lack access to evidence-based treatments. Community lay-therapists are a promising solution for the global mental health field. However, in spite of results from randomized-control trials, no research to-date has examined the external validity of community-led lay-therapist effectiveness. In this exploratory study, longitudinal data at three time points were collected from 28 Arabic-speaking displaced persons (nineteen women and nine men, ages 18-57) seeking mental health services from the Jiyan Foundation: a non-profit founded and based in Kurdish Iraq. Lay therapists trained in evidence-based treatments upon being hired operated largely independently of supervision from foreign clinicians. Participants in weekly psychotherapy completed the Posttraumatic Stress Checklist (PCL-5) and the Psychological Health Questionnaire (PHQ-9) at baseline, one month, and three months, as well as a modified measure assessing traumatic exposure, purpose-in-life, and a modified Afghan Daily Stressors Scale at baseline to assess for moderators of change over time.

ELIGIBILITY:
Inclusion Criteria:

* Must speak Arabic fluently; must be seeking mental health services at the Jiyan Foundation

Exclusion Criteria:

* No Arabic proficiency; under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were 18-years-or-older Arabic speakers displaced from their homes in either Central/Southern Iraq or Syria and now residing in Kurdish Iraq and seeking treatment for mental health difficulties.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms | 3 months
  Measured by the PCL-5
Depression Symptoms | 3 months
  Measured by the PHQ-9

CONTACTS AND LOCATIONS:
Locations (1):
- Jiyan Foundation for Human Rights, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Dataset is available with participant answers, but original forms are not to be shared as some personal information was written in notes (i.e. names)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available for two years after reporting and by request following.
Access Criteria: Data is publicly available at OSF for download, or can be requested by contacting blackwell@unm.edu